CLINICAL TRIAL: NCT03523884
Title: Development of A Technology-Enabled Intervention for Musculoskeletal Health: The Effectiveness of Technology-enabled Exercise Program in Firefighters With Shoulder Pain. A Randomized Controlled Trial.
Brief Title: Effectiveness of Technology-enabled Exercise Program in Firefighters With Shoulder Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UWO Firefighters 2018
Record Dates: First submitted 2018-04-11; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Educational Status; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Program plus Education. (Experimental): Rotator cuff stretching and strengthening exercises outlined in the American Academy of Orthopedic Surgeons (AAOS) guidelines on management of rotator cuff problems.
  Interventions: Other: Exercise Program plus Education; Other: Educational Program (EP).
- Educational Program (EP). (Active Comparator): An information sheet form AAOS, outlining the anatomy, description, causes, symptoms, examination and imaging tests performed on individuals with shoulder conditions
  Interventions: Other: Educational Program (EP).

INTERVENTIONS:
Other: Exercise Program plus Education — Rotator cuff exercises outlined in the American Academy of Orthopedic Surgeons (AAOS) guidelines on management of rotator cuff problems.
  Other Names: Exercise and Education
  Arms: Exercise Program plus Education.
Other: Educational Program (EP). — An information sheet form AAOS, outlining the anatomy, description, causes, symptoms, examination and imaging tests performed on individuals with shoulder conditions
  Other Names: Education.

SUMMARY:
To assess if a technology-enabled Exercise program plus Education (TEEP + E) is more effective than Education program (EP) alone, in providing better outcomes (quality of life, at-work disability and productivity loss, firefighters' perception, adherence, overall improvement/deterioration) in firefighters with shoulder pain, at 3-, 6-and 12-month follow ups.

ELIGIBILITY:
Inclusion Criteria:

* Active duty firefighters aged 18 to 100 years, with shoulder pain.
* Do not permanently use strong pain medications.
* Able to understand spoken and written English.
* Access to computer, internet and telecommunications application software (Skype).

Exclusion Criteria:

* Firefighters who have had shoulder related surgeries in the last 6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Firefighter Work Limitation Questionnaire | 3-months
  at-work disability and productivity loss
Firefighter Work Limitation Questionnaire | 6-months
  at-work disability and productivity loss
Firefighter Work Limitation Questionnaire | 12-months
  at-work disability and productivity loss
Short- Western Ontario Rotator Cuff Index | 3-months
  Quality of life
Short- Western Ontario Rotator Cuff Index | 6-months
  Quality of life
Short- Western Ontario Rotator Cuff Index | 12-months
  Quality of life

SECONDARY OUTCOMES:
Single Assessment Numeric Evaluation | 3-, 6- and 12-months
  Patient's perception of the condition
Number of days lost | 3-, 6- and 12-months
  Work days lost due to the condition
Therapy Adherence Assessment Tool | 3-, 6- and 12-months
  Exercise adherence
Global Rating of Change Scale | 6- and 12-months
  To quantify a patient's improvement or deterioration over time
Adverse Effects | 3-, 6- and 12-months
  Have you experienced any exercise-induced pain

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Study Chair — Western University, jmacderm@uwo.ca, 519 661 2111 x (88912)
Locations (1):
- Hamilton Fire Station, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No